CLINICAL TRIAL: NCT01557803
Title: Prediction and Pathogenesis of the Immune Reconstitution Inflammatory Syndrome in Lambaréné, Gabon
Brief Title: Prediction and Pathogenesis of the Immune Reconstitution Inflammatory Syndrome
Acronym: IRIS
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: University Hospital Tuebingen (Other); Albert Schweitzer Hospital (Other)
Responsible Party: Principal Investigator, S. Janssen, MD, MSc, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: MRU-HAS 006/2012; NCT01549821 (obsolete NCT alias)
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Immune Reconstitution Inflammatory Syndrome; Opportunistic Infections
Keywords: Immune reconstitution inflammatory syndrome; Biomarkers; HIV; ART; predictive factors; epidemiological pattern; Gabon
MeSH Terms: conditions — Immune Reconstitution Inflammatory Syndrome; Opportunistic Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, Paxgene RNA tubes and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Starting ART: Adult patients starting anti retroviral therapy for the first time

SUMMARY:
The objective of this project is to determine clinical and biological predictors of Immune Reconstitution Inflammatory Syndrome (IRIS) occurrence in HIV infected patients who are started on antiretroviral therapy (ART), and to obtain more insight into the pathogenesis of this syndrome. The investigators will prospectively study HIV infected patients in Sub Saharan Africa who will be initiated on ART and are at risk to develop IRIS in all its different appearances. In these patients, the investigators will assess the value of clinical features and plasma biomarkers to predict IRIS, and the investigators will obtain insight into which inflammatory pathways become activated during IRIS. This project will provide novel knowledge about this clinically highly relevant healthcare problem in a resource poor setting, namely in Lambaréné, Gabon, in the Central African rainforest belt. In Gabon little research has been done in the field of HIV. The epidemiological pattern of IRIS in Gabon will be described. Promising putative plasma biomarkers will be validated for their use in daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Informed consent
* ART naive

Exclusion Criteria:

* No informed consent
* History of ART use
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult HIV patients starting anti retroviral therapy for the first time
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
IRIS | 12 months
  Development of immune reconstitution inflammatory syndrome

SECONDARY OUTCOMES:
Time to IRIS | 12 months
  Time to development of immune reconstitution inflammatory syndrome

CONTACTS AND LOCATIONS:
Overall Officials: MP Grobusch, MD, MSc, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Medical Research Unit - Albert Schweitzer Hospital, Lambaréné, Moyen Ogoué, Gabon